CLINICAL TRIAL: NCT05895708
Title: Effect of Specific Postural Corrective Exercises on EMG Activity of Masticatory and Cervical Muscles in Patients With Forward Head Posture
Brief Title: Effect of Specific Postural Corrective Exercises on EMG Activity in Patients With Forward Head Posture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beirut Arab University (Other)
Responsible Party: Principal Investigator, Rami Abbas, Associate Prof of Physical Therapy Assistant Dean Faculty of Health Sciences, Beirut Arab University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Forward Head Posture
Record Dates: First submitted 2023-04-03; First posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Forward Head Posture

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Specified strengthening and stretching (Experimental): The program consisted of two strengthening (deep cervical flexors and shoulder retractors) and two stretching (cervical extensors and pectoral muscles) exercises based on Harman and Mostafa et al's approach. This exercise program will be repeated 4 times per week for 10 weeks, and each session lasted for 30 minutes.
  Interventions: Other: Specific strengthening and stretching exercise
- General Exercise group (Sham Comparator): The program will consist of regular general postural exercises such as postural awareness exercises as well as general strengthening exercises such as range of motion exercises for the upper quadrant. The program will also be repeated 4 times per week for 10 weeks, with each session lasting 30 minutes
  Interventions: Other: General Exercise

INTERVENTIONS:
Other: Specific strengthening and stretching exercise — The program consisted of two strengthening (deep cervical flexors and shoulder retractors) and two stretching (cervical extensors and pectoral muscles) exercises based on Harman and Mostafa et al's approach. This exercise program will be repeated 4 times per week for 10 weeks, and each session lasted for 30 minutes.
  Other Names: Forward head correction
  Arms: Specified strengthening and stretching
Other: General Exercise — The program will consist of regular general postural exercises such as postural awareness exercises as well as general strengthening exercises such as range of motion exercises for the upper quadrant. The program will also be repeated 4 times per week for 10 weeks, with each session lasting 30 minutes
  Arms: General Exercise group

SUMMARY:
This study investigates the effects of specific corrective exercises on EMG of masticatory and cervical muscles in patients with forward head posture. The study's design will be a prospective, double- blinded, randomized controlled trial. The participants will be randomly allocated to one of two groups: the exercise group and the control group. The training groups will perform a program consisting of two strengthening (deep cervical flexors and shoulder retractors) and two stretchings (cervical extensors and pectoral muscles) exercises. This exercise program will be repeated 4 times per week for 10 weeks, and each session lasted 30 minutes.

The pre/post assessment of forward head posture will measure by using craniovertebral angle CVA. While the muscle activity EMG of the masseter, temporalis, splenius, upper trapezius, and SCM will measure pre and post-assessment using a biopic data acquisition system. There will be a high significance increase (p-value 0.000) between the pre-and-post CVA between the training groups and the control. And there will be a significant decrease in EMG of the masseter, temporalis, splenius, upper trapezius, and SCM across exercise groups compared to the control. As per the results and analysis, specific postural corrective exercises effectively decrease the EMG of masticatory and cervical muscles in patients with forward head postures.

DETAILED DESCRIPTION:
Forward head posture (FHD) is a common habitual faulty posture exists in the surrounding that can alter the resting position of the mandible and may affect the masticatory muscle activity.

The aim of this study is to investigate the effect of postural correction on masticatory and cervical muscle activity and mandibular opening in forward-head posture patients.

Materials and Methods:

* Cranio-vertebral angle measurement CVA
* EMG activity of masseter, temporalis, splenius, upper trapezius and SCM

BAU - Institutional Review Board (Form H-II) | BEIRUT ARAB UNIVERSITY

-Electrodes will be placed on the muscle belly parallel to the direction of muscle fibers. The distance between the two electrodes was 2 cm. The subjects will be instructed to complete maximum voluntary contraction (MVC) of clenching the teeth for 3 s and repeating twice. The average of the two trials of MVC will be used for further analysis. The subjects will be seated comfortably in a chair (---cm height).

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Age between 18-40
* Patient with forward head posture, CVA less than 48-50.
* Patient suffer from temporomandibular joint disorder
* No other treatment, such as medication, physical therapy, and joint injection, in the past 2 weeks

Exclusion Criteria:

* Previous history of TMG subluxation or dislocation that may interfere with the opening of the mouth
* Neck pain which may affect the head and neck posture;
* Head or neck trauma
* Class II or III malocclusion
* Posture disorder caused by abnormal curvature of spine; rheumatic disease; haemorrhagic disease, etc.; and
* Lateral deviation of mandible

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-06-15 (Estimated); Primary Completion 2023-09-20 (Estimated); Study Completion 2023-09-20 (Estimated)

PRIMARY OUTCOMES:
EMG activity | 12 weeks
  Electrodes will be placed on the muscle belly parallel to the direction of muscle fibers. The distance between the two electrodes was 2 cm.
  The subjects will be instructed to complete maximum voluntary contraction (MVC) of clenching the teeth for a period of 3 s and repeated twice. The average of the two trials of MVC will be used for further analysis. The subjects will be seated comfortably in a chair (---cm height).

OTHER OUTCOMES:
craniovertebral angle | 12 weeks
  Forward head posture will be assess by the craniovertebral angle, one of the most reliable tool for evaluating the FHP.
  The examiner takes 2 lateral photographs of the subject in standing position, according to Shaghayegh fard et al.
  A digital camera will be positioned on a tripod at a distance of 0.8m from the subject at shoulder height. Two land mark will be taken, the spinous process of C7 and the tragus of ear. A horizontal line will be drawn passing through C7 making a right angle with the vertical. Then, the angle between the line connecting C7 spinous process with the tragus of the ear and the horizontal line.

CONTACTS AND LOCATIONS:
Overall Officials: ahmed el melhat, professor, Study Director — Beirut Arab University
Locations (1):
- Physical therapy outpatient clinic, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No
Any study records that identify patient will be kept confidential. The records from the participation may be reviewed by people responsible for making sure that research is done properly, including members of the BAU Institutional Review Board. All of these people are required to keep their identities confidential. Otherwise, records that identify patients will be available only to people working on the study.
  • The investigators will use a code of numbers and alphabets rather than participants' names on data sheets, keeping records in a safe place.

REFERENCES:
- [Background] Shaghayegh Fard B, Ahmadi A, Maroufi N, Sarrafzadeh J. Evaluation of forward head posture in sitting and standing positions. Eur Spine J. 2016 Nov;25(11):3577-3582. doi: 10.1007/s00586-015-4254-x. Epub 2015 Oct 17. PMID 26476717
- [Background] Zabihhosseinian M, Holmes MW, Ferguson B, Murphy B. Neck muscle fatigue alters the cervical flexion relaxation ratio in sub-clinical neck pain patients. Clin Biomech (Bristol). 2015 Jun;30(5):397-404. doi: 10.1016/j.clinbiomech.2015.03.020. Epub 2015 Mar 27. PMID 25843481
- [Background] Lee KJ, Han HY, Cheon SH, Park SH, Yong MS. The effect of forward head posture on muscle activity during neck protraction and retraction. J Phys Ther Sci. 2015 Mar;27(3):977-9. doi: 10.1589/jpts.27.977. Epub 2015 Mar 31. PMID 25931773
- [Background] Quek J, Pua YH, Clark RA, Bryant AL. Effects of thoracic kyphosis and forward head posture on cervical range of motion in older adults. Man Ther. 2013 Feb;18(1):65-71. doi: 10.1016/j.math.2012.07.005. Epub 2012 Sep 5. PMID 22959228
- [Background] Lee SM, Lee CH, O'Sullivan D, Jung JH, Park JJ. Clinical effectiveness of a Pilates treatment for forward head posture. J Phys Ther Sci. 2016 Jul;28(7):2009-13. doi: 10.1589/jpts.28.2009. Epub 2016 Jul 29. PMID 27512253
- [Background] Kim SD. Effects of yoga exercises for headaches: a systematic review of randomized controlled trials. J Phys Ther Sci. 2015 Jul;27(7):2377-80. doi: 10.1589/jpts.27.2377. Epub 2015 Jul 22. PMID 26311986